CLINICAL TRIAL: NCT05993715
Title: Influence of Nitrate Supplementation on Motor Unit Activity During Recovery Following a Sustained Ischemic Contraction.
Brief Title: Nitrate Supplementation on Motor Unit Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Ozcan Esen, Assistant Professor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 5951
Record Dates: First submitted 2023-06-20; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Dietary Supplements; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Supplements were allocated in a randomised order and double-blind design by an independent technician who had no further involvement in this study. The randomization and blinding were held until the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate supplementation (Experimental): 2 × 70 mL/day shots of concentrate nitrae-rich (~12.8 mmol/day NO3-) beetroot juice. Two shots were supplemented for 5 days; one each morning (~9 am) and one each evening (~9 pm) except for the day of the experimental trial when both shots were taken together 2.5 h before the experimental trial.
  Interventions: Dietary Supplement: Nitrate supplementation
- Placebo supplementation (Placebo Comparator): 2 × 70 mL/day shots of concentrate nitrate-depleted (~0.08 mmol/day NO3-) beetroot juice. Two shots were supplemented for 5 days; one each morning (~9 am) and one each evening (~9 pm) except for the day of the experimental trial when both shots were taken together 2.5 h before the experimental trial.
  Interventions: Dietary Supplement: Placebo supplementtaion

INTERVENTIONS:
Dietary Supplement: Nitrate supplementation — Participants ingested 2 × 70 mL/day shots of concentrate nitrate-rich (~12.8 mmol/day nitrate) or nitrate-depleted (~0.08 mmol/day nitrite) beetroot juice (Beet It, James White Drinks Ltd., Ipswich, UK). Two shots were supplemented for 5 days; one each morning (~9 am) and one each evening (~9 pm) except for the day of the experimental trial when both shots were taken together 2.5 h before the experimental trial.
  Arms: Nitrate supplementation
Dietary Supplement: Placebo supplementtaion — 2 × 70 mL/day shots of concentrate nitrate-depleted (~0.08 mmol/day NO3-) beetroot juice. Two shots were supplemented for 5 days; one each morning (~9 am) and one each evening (~9 pm) except for the day of the experimental trial when both shots were taken together 2.5 h before the experimental trial.
  Arms: Placebo supplementation

SUMMARY:
This study aimed to assess if nitrate supplementation influence motor unit (MU) activity following a sustained ischemic contraction and whether this is affected by blood flow restriction (BFR) during the recovery period. Fourteen male participants (mean ± SD, 25 ± 6 years) completed two experimental trials following 5-days of supplementation with either nitrate-rich (NIT) or nitrate-depleted (PLA) beetroot juice in a randomized, double-blinded, cross-over design. Intramuscular electromyography was used to assess MU potential (MUP) size and firing rates (MUFR) during a submaximal (25% MVC) sustained isometric contraction with BFR. These variables were also assessed during a 90 s recovery period with the first half completed with, and the second half completed without, BFR. Nitrate supplementation can expedite the recovery of MUP duration following a sustained ischemic contraction in healthy adults. These novel observations improve understanding of the effects of nitrate on the recovery of neuromuscular function post-exercise and might have implications for recovery of muscle contractile function.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 - 30 years
* free from known respiratory insufficiency, cardiovascular disease and neuro-musculo-skeletal problems at present or in the preceding 6 months.
* having at least 5 years competitively (team) sport experience.

Exclusion Criteria:

* having cardiovascular disease, neuromuscular disease and any lower limb injury and treatment for chronic respiratory complaints.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma Nitrite Level | Pre-exercise
  concentration [nmol]
Motor Unit Activity | Pre-exercise, post-exercise, recovery (45 s)
  Duration (ms), area (uV.ms), firing rate (Hz)

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esen O, Bailey SJ, Stashuk DW, Howatson G, Goodall S. Influence of nitrate supplementation on motor unit activity during recovery following a sustained ischemic contraction in recreationally active young males. Eur J Nutr. 2024 Sep;63(6):2379-2387. doi: 10.1007/s00394-024-03440-9. Epub 2024 May 29. PMID 38809323